CLINICAL TRIAL: NCT05993624
Title: The Effect of Exergame Games on Kinesiophobia, Balance, Lower Extremity Muscle Strength, Depression and Cognitive Function in Geriatric Individuals With Kinesiophobia
Brief Title: The Effect of Exergame Games on Geriatric Individuals With Kinesiophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Sever, PhD, PT, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELMİRAHASRET
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Geriatric; Kinesiophobia
Keywords: geriatrics; kinesiophobia; virtual reality; video based game; Xbox 360 KinectTM
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation Group (Other): Participants in the study played 30-minute exergame games once a week for 8 weeks and rehabilitation was applied. Before starting the application, the participants were given a demographic information form, Tampa kinesiophobia scale for kinesiophobia, BeCure balance assessment system for balance measurement, geriatric depression scale-short form for depression, mini-mental state test for cognitive functions, and lower extremity functional strength. and 5 times the risk of falling. lifting test was performed. These tests were repeated at the end of 8 sessions and before and after values were measured.
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — The BeCure Balance Assessment System protocol used in this study; It was planned to determine the amount of change in the center of gravity in the x and y axes and the position of the center of gravity of the body with images during standing and balancing for 15 seconds on the board with eyes open. In order to support the balanced development of the participants with the Becure system; Balance surfing, balance adventure, balance bowling and traffic games were played. uBall, gates, smartclean and SmartBubblePop games with Kinect for the upper extremity; KneeUp game was played on the lower extremity.

SUMMARY:
The study included 15 geriatric individuals over the age of 65 staying in Kızılay Zeynep Nedim Oyvar Nursing Home and Elderly Nursing Home. Participants in the study were rehabilitated by playing exergame games with Xbox 360 KinectTM for 30 minutes once a week for 8 weeks. Before starting the application, the participants were given a demographic information form, Tampa kinesiophobia scale for kinesiophobia, Nintendo Wii balance platform and basic balance game for balance measurement, geriatric depression scale-short form for depression, cognitive functions, and mini-mental state test for the lower extremities. functional strength and risk of falling. The shuttle test was applied 5 times. These tests will be repeated at the end of 8 sessions and before and after values were measured. As a result of the analysis, the effects of Xbox 360 KinectTM games on kinesiophobia, balance, lower extremity muscle strength, depression, and cognitive functions in geriatric individuals with kinesiophobia were investigated.

DETAILED DESCRIPTION:
15 geriatric individuals over 65 years old living in Kızılay Zeynep Nedim Oyvar Nursing Home and Elderly Care Center were included in the study. The ethics committee of Istanbul Gedik University Ethics Committee, dated 17/01/2023 and numbered E-56365223-050.01.04-2023.137548.27-433, was accepted. A consent form was signed by geriatric individuals who met the conditions of this study. Participants participating in the study played 30 minutes of exergame games once a week for 8 weeks and rehabilitation was applied. Before starting the application, participants were given a demographic information form, Tampa kinesiophobia scale for kinesiophobia, BeCure balance assessment system for balance measurement, geriatric depression scale-short form for depression, mini-mental state test for cognitive functions, and lower extremity functional strength and risk of falling 5 times. lift test was applied. These tests were repeated at the end of 8 sessions and before and after values were measured.

ELIGIBILITY:
Inclusion Criteria:

* Getting 38 or higher on the Tampa Kinesiophobia Scale
* Getting a Mini Mental State Test Score of 20 and above
* Being physically competent to apply the scales to be used
* Being 65 years or older
* Volunteering to work

Exclusion Criteria:

* Having a mental and psychiatric problem diagnosed by a physician
* Having a serious neurological and orthopedic problem diagnosed by a physician
* Having serious hearing and vision problems
* Having uncontrolled diabetes and hypertension
* Using a walking device other than a cane (crutches, walkers, etc.)
* Drug use that increases the risk of falling (to be determined by the information obtained from nurses and physiotherapists working in nursing homes)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | 8 weeks
  It measures fear of movement and fear of re-injury. It was used to evaluate the development of fear of movement after treatment. A 4-point Likert scoring (1= I strongly disagree, 4= I totally agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. The person gets a total score between 17-68. A high score on the scale indicates that kinesiophobia is also high.
BeCure Balance Evaluation System | 8 weeks
  The BeCure Balance Assessment System protocol used in this study; It was planned to determine the amount of change in the center of gravity in the x and y axes and the position of the body center of gravity during standing balance on the board for 15 seconds with eyes open, with images.

SECONDARY OUTCOMES:
Geriatric Depression Scale- Short Form | 8 weeks
  It consists of 15 questions questioning the mood in the last week. This short form consists of 15 questions questioning the mood of the patient. The answers are given according to the feelings in the last week; The answers are "yes" or "no", just like in the long form, and 1 point is given for "yes" or "no" answers depending on the question. A score of 0-4 indicates no depression, 5-8 indicates mild depression, 9-11 indicates moderate depression, and a score of 12-15 indicates severe depression.
Mini Mental State Test | 8 weeks
  Cognitive testing of the elderly, especially the elderly with delirium and/or dementia.A minimum of 0 and a maximum of 30 points can be obtained from this test. It is thought that the higher the score, the worse the mental state of the individual.
5 Times Sit Up Test | 8 weeks
  It is a test used to evaluate the functional strength, balance and fall risk of the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru SEVER, Lecturer, Study Director — Department of Physiotherapy & Rehabilitation
Locations (1):
- Kızılay Zeynep Nedim Oyvar Nursing Home and Elderly Care Center, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No